CLINICAL TRIAL: NCT03317717
Title: Phase 1 Study to Determine the Pharmacodynamic and Safety of MEDITOXIN®(Clostridium Botulinum Toxin Type A) in Healthy Male Volunteers
Brief Title: Pharmacodynamic and Safety of MEDITOXIN® in Healthy Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Medy-Tox (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: MT01-KR17EDB107
Record Dates: First submitted 2017-10-18; First posted 2017-10-23 (Actual); Last update posted 2019-03-27 (Actual); Status verified 2019-03

CONDITIONS: Healthy
MeSH Terms: interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- botulinum toxin 2U (Experimental)
  Interventions: Drug: Meditoxin; Drug: Botox
- botulinum toxin 5U (Experimental)
  Interventions: Drug: Meditoxin; Drug: Botox
- botulinum toxin 10U (Experimental)
  Interventions: Drug: Meditoxin; Drug: Botox
- botulinum toxin 20U (Experimental)
  Interventions: Drug: Meditoxin; Drug: Botox
- botulinum toxin 30U (Experimental)
  Interventions: Drug: Meditoxin; Drug: Botox

INTERVENTIONS:
Drug: Meditoxin — injection of MEDITOXIN into EDB muscle of one foot and BOTOX into the same muscle of contralateral foot in equal doses
Drug: Botox — injection of MEDITOXIN into EDB muscle of one foot and BOTOX into the same muscle of contralateral foot in equal doses

SUMMARY:
This study will determine the pharmacodynamic and safety of MEDITOXIN® in healthy male volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Male adults aged between 20 and 45
* Satisfying baseline nerve conduction criteria in below at screening visit CMAP M-wave amplitude of EDB ≥ 4.0mV CMAP M-wave amplitude of AH ≥ 5.0mV CMAP M-wave amplitude of ADQ ≥ 5.0mV

Exclusion Criteria:

* Have history of childhood botulism
* Have a pacemaker or any other heart device
* Have peripheral neuropathy or accessary peroneal nerve
* Have history of lower limb myotomy or denervation surgery

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2017-10-12 (Actual); Primary Completion 2018-01-30 (Actual); Study Completion 2018-01-30 (Actual)

PRIMARY OUTCOMES:
CMAP(Compound Muscle Action Potential) amplitude of the EDB(Extensor Digitorum Brevis) muscle | day 14, 30, 60, 90
  percentage reduction of CMAP(Compound Muscle Action Potential) amplitude of the EDB(Extensor Digitorum Brevis) muscle from baseline

CONTACTS AND LOCATIONS:
Locations (1):
- The Catholic University of Korea, St. Paul's Hospital, Seoul, South Korea